CLINICAL TRIAL: NCT06306807
Title: Investigation of the Effectiveness of Proprioceptive Neuromuscular Facilitation Techniques in Text Neck Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Meltem Kaya, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AtlasUmkaya02
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Neck Muscle Issue
Keywords: Text Neck Syndrome; Neck Pain; Range of Motion; Posture; Disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group underwent the exercise program including active cervical range of motion, strengthening, and posture correction exercises for 6 weeks, 3 days a week, once a day for 10 repetitions. Active cervical range of motion exercise program consists of the general range of movement for flexors, extensors, both sides flexors, and rotator neck muscles. Strengthening exercises were planned for weak, lengthened, inhibited muscles. Ergonomic modifications while using a smartphone were taught. Additionally, participants in the experimental group were included in a PNF exercise program to be applied by a physiotherapist 3 days a week for 6 weeks. The contract-relax technique for the neck extension pattern and the replication technique for the scapular posterior elevation pattern were used.
  Interventions: Other: Exercise program including active cervical range of motion, strengthening, and posture correction exercises and ergonomic modifications; Other: PNF exercise program
- Control Group (Active Comparator): Participants in the experimental group underwent the exercise program including active cervical range of motion, strengthening, and posture correction exercises for 6 weeks, 3 days a week, once a day for 10 repetitions. Active cervical range of motion exercise program consists of the general range of movement for flexors, extensors, both sides flexors, and rotator neck muscles. Strengthening exercises were planned for weak, lengthened, inhibited muscles. Ergonomic modifications while using a smartphone were taught.
  Interventions: Other: Exercise program including active cervical range of motion, strengthening, and posture correction exercises and ergonomic modifications

INTERVENTIONS:
Other: Exercise program including active cervical range of motion, strengthening, and posture correction exercises and ergonomic modifications — Active cervical range of motion exercise program consists of the general range of movement for flexors, extensors, both sides flexors, and rotator neck muscles. Participants were instructed to perform exercises in a sitting position, but they were allowed to perform exercises in supine and prone lying if they had problems with sitting position. Strengthening exercises were planned for weak, lengthened, inhibited muscles e.g. Longus colli, and longus capitis. Chin tucks, chin tucks against gravity, and chin nod exercises were selected. Ergonomic modifications while using a smartphone were taught such as taking breaks and changing positions frequently while using a smartphone, avoiding cradling the phone between your ear and shoulder, choosing a smartphone that fits your hands properly, holding the smartphone near chest level rather than waist level, and using features including predictive text or auto-complete tools
Other: PNF exercise program — The contract-relax technique for the neck extension pattern and the replication technique for the scapular posterior elevation pattern were used.
  Arms: Experimental Group

SUMMARY:
Smartphones and tablets are increasingly widespread mobile technological devices used for many purposes such as communication, transportation, entertainment, education and security. Increasing use of mobile technology leads to various symptoms such as insomnia, difficulty concentrating and anxiety, especially musculoskeletal problems. "Text neck" is a musculoskeletal problem seen in individuals who use smartphones and tablets for a long time due to increased head and neck flexion posture. It causes neck, back, shoulder, and head pain, insomnia, tingling and numbness in the hands. Implementation of exercise programs for both preventive and therapeutic purposes is one of the main goals in this picture dominated by posture and pain problems. Proprioceptive neuromuscular facilitation (PNF) treatment technique; In the 1940s by H. Kabat and M. Knott, PNF was expressed as a means of facilitating neuromuscular responses by stimulation of proprioceptors. It is stated that it increases joint stabilization, strength, normal range of motion, endurance and circulation and is effective in improving coordination. Although PNF techniques have been used for different spinal problems, there is no study investigating PNF techniques in text neck syndrome. The study was aimed to compare the effect of a method including muscle relaxation in the anterior elevation direction and repetition techniques in the posterior depression direction from PNF neck patterns on pain intensity, neck normal range of motion, neck muscle endurance, posture and functionality in individuals with text neck syndrome with another method including ergonomic adjustments and simple cervical exercises recommended in the literature to be included in standard treatment.

DETAILED DESCRIPTION:
Smartphones and tablets are increasingly widespread mobile technological devices used for many purposes such as communication, transportation, entertainment, education and security. Increasing use of mobile technology leads to various symptoms such as insomnia, difficulty concentrating and anxiety, especially musculoskeletal problems. "Text neck" is a musculoskeletal problem seen in individuals who use smartphones and tablets for a long time due to increased head and neck flexion posture. It causes neck, back, shoulder, and head pain, insomnia, tingling and numbness in the hands. Implementation of exercise programs for both preventive and therapeutic purposes is one of the main goals in this picture dominated by posture and pain problems. Proprioceptive neuromuscular facilitation (PNF) treatment technique; In the 1940s by H. Kabat and M. Knott, PNF was expressed as a means of facilitating neuromuscular responses by stimulation of proprioceptors. It is stated that it increases joint stabilization, strength, normal range of motion, endurance and circulation and is effective in improving coordination. Although PNF techniques have been used for different spinal problems, there is no study investigating PNF techniques in text neck syndrome. The study was aimed to compare the effect of a method including muscle relaxation in the anterior elevation direction and repetition techniques in the posterior depression direction from PNF neck patterns on pain intensity, neck normal range of motion, neck muscle endurance, posture and functionality in individuals with text neck syndrome with another method including ergonomic adjustments and simple cervical exercises recommended in the literature to be included in standard treatment. Our study is planned as a randomized controlled, prospective, single-blind case-control study. Demographic and clinical information of all participants to be included in the study will be recorded with the "Demographic and Clinical Information Form". Neck pain will be assessed by visual analog scale (VAS), cervical joint normal range of motion will be assessed by cervical flexion, cervical extension, cervical lateral flexion and cervical rotation normal range of motion measurements, neck muscle endurance will be assessed by neck flexor and extensor muscle endurance tests, posture will be assessed by New York Posture Evaluation Scale and functionality will be assessed by Neck Disability Index.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year of using a smartphone
* using smartphones>4 hours per day, having recurrent neck pain which is increased by sustained posture and feeling of stiffness on turning the head and neck after long usages
* be able to read written and understand spoken language and willing to participate were included.

Exclusion Criteria:

* Subjects with spinal infections or inflammatory disorders
* a history of neck surgery, trauma, torticollis, scoliosis, malignancies, pregnancy, diagnosed disc prolapse, stenosis, herniation, spondylolisthesis, osteoporosis
* currently continuing or participating in a regular exercise program
* unable to perform tests or exercises because of diagnosed comorbidities or presently undergoing medication or physical therapy treatments

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 6 weeks
  The neck pain score was measured using the visual analog scale. The VAS is a subjective scoring method for recording the degree of present pain from 0 (no pain) to 10 (the most severe pain ever experienced) on a 10-cm scale. The minimum clinical important difference (MCID) for VAS is 1.4 cm (on a 10 cm scale)
Cervical range of motion | 6 weeks
  Active cervical range of motion was measured in all directions with a plastic universal goniometer. Participants were instructed to sit upright while securing their thoracic area to a chair to assess their cervical range of motion. They were then directed to perform a series of standard movements: flexion, extension, left-right lateral flexion, and left-right rotation. Three consecutive measurements were obtained and the average value was recorded as degree. Before measurements, all participants were encouraged to perform each neck movement to the end range to familiarize themselves with the testing method and to reduce the creep.
Neck flexor-extensor muscle endurance test | 6 weeks
  The neck flexor muscle endurance test was performed in the supine and crook lying position. The participant lifted the head and neck until the head was approximately 2.5 cm off the plinth. The "hold your head up" command was given. The test was stopped if the participant's head touched the investigator's hand for over one second. Holding time was recorded in seconds with a stopwatch. The neck extensor muscle endurance test was performed in the prone position. The participant was asked to retract the chin and hold the head steady horizontally. The test was stopped if the subject could not maintain the head in a horizontal position. The endurance time was measured in seconds by stopwatch
Posture | 6 weeks
  The evaluation of posture involved using the New York Posture Rating Chart (NYPR), a cost-effective, easily applicable method commonly employed for subjective postural assessment in clinical settings. This chart allows for the assessment of 13 body areas, based on the idea that posture reflects the body's alignment and its various segments.
Disability | 6 weeks
  The assessment of disability relied on the Neck Disability Index (NDI), comprising a self-reported scale of 10 items. Each item addresses various complaints related to neck pain, primarily focusing on limitations in activities of daily living. Each item is represented by six different statements, graded on a scale from 0 to 5, where 0 denotes no disability and 5 signifies the most severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No